CLINICAL TRIAL: NCT05348317
Title: Using Telehealth to Expand Treatment Access for Veterans With Opioid Use Disorder (CDA 18-008)
Brief Title: Developing a Telehealth Model to Improve Treatment Access for Rural Veterans With Substance Use Disorders
Acronym: VetReach
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Ann Arbor Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX 22-007; PROJ-03672 (Other: VA Ann Arbor Healthcare System)
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Substance Use; Substance Use Disorders; Substance Dependence; Veterans
Keywords: Telehealth; Motivational Interviewing; Cognitive Behavioral Therapy; Rural Health
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MI-CBT Teletx (Experimental): The intervention consists of an initial 30-60 min phone-delivered Engagement session that focuses on MI to help participants build self-efficacy and motivation to engage and to empower them to plan change and use Elicit-Provide-Elicit (EPE) to address treatment barriers (e.g., stigma, appeal, accessibility). Participants will then complete up to 8 ~50 minute Teletx weekly sessions via videoconference (or phone if needed). The intervention is highly patient-centered, by meeting and assessing patients where they are including in their unique context (i.e. rural community), helping them identify reasons and motivations for change, and centered around their goals (e.g. substance use reduction or abstinence).
  Interventions: Behavioral: VetReach

INTERVENTIONS:
Behavioral: VetReach — Telehealth-delivered MI-CBT substance use disorder care model

SUMMARY:
This project will pilot-test and obtain stakeholder input on a telehealth-delivered substance use disorder (SUD) care model (with initial engagement and ongoing MI-CBT treatment) with the goal of increasing treatment utilization and improving outcomes for rural and non-rural Veterans with SUDs.

ELIGIBILITY:
Inclusion Criteria:

* Veteran patients at the Ann Arbor VA Healthcare System
* Diagnostic and Statistical Manual of Mental Disorders (DSM-5) SUD diagnosis and/or substance use on average of 2 days a week over the past month
* Telephone access
* Able to provide informed consent

Exclusion Criteria:

* Receiving SUD psychotherapy
* Inability to speak or understand English
* Substantial mental health instability or conditions that preclude informed consent (e.g., acute psychosis, cognitive deficits) or understanding of assessment or program content
* Prior alcohol withdrawal seizures or delirium tremens

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention (engagement) | 8 weeks
  Percent (%) of participants engaging in the intervention (at least 3 completed sessions)
Acceptability of the telehealth intervention | 2 months
  Study-specific acceptability rating completed by participants (% with a positive rating, higher % is better)

OTHER OUTCOMES:
Change in substance consumption | baseline, 8 weeks post-baseline
  Substance use/consumption will be assessed using the 30-day Timeline Follow-Back (TLFB). The TLFB will capture information on the frequency and quantity of substance use, with total consumption calculated.
Change in frequency of substance use as reported on the Timeline Follow-Back (TLFB) | baseline, 8 weeks post-baseline
  Based on frequency and quantity, higher scores indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lewei Lin, MD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT05348317/ICF_000.pdf